CLINICAL TRIAL: NCT06543069
Title: A Single-Arm, Phase II Clinical Study of Sintilimab and Bevacizumab Combined With Pemetrexed and Cisplatin for Unresectable Malignant Peritoneal Mesothelioma
Brief Title: Sintilimab, Bevacizumab, Pemetrexed, and Cisplatin for Unresectable MPeM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4469
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Malignant Peritoneal Mesothelioma, Advanced
Keywords: Sintilimab; Bevacizumab; Pemetrexed; Cisplatin; Malignant Peritoneal Mesothelioma
MeSH Terms: interventions — sintilimab; Bevacizumab; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Sintilimab and Bevacizumab Combined with Pemetrexed and Cisplatin
  Interventions: Drug: Sintilimab, Bevacizumab , Pemetrexed , Cisplatin

INTERVENTIONS:
Drug: Sintilimab, Bevacizumab , Pemetrexed , Cisplatin — Sintilimab: 200mg, bevacizumab: 7.5mg/kg, pemetrexed: 500mg/m2, cisplatin: 75mg /m2, Q3w. Tumor assessments will be performed every two cycles according to RECIST 1.1 criteria. After 6 cycles, maintenance therapy with sintilimab, bevacizumab, and pemetrexed will continue until disease progression or unacceptable toxicity occurs.
  Other Names: Sintilimab+Bevacizumab+Pemetrexed+ Cisplatin

SUMMARY:
To explore the efficacy and safety of sintilimab, bevacizumab combined with pemetrexed and cisplatin in the treatment of malignant peritoneal mesothelioma, and to explore the biomarkers related to efficacy or safety.

DETAILED DESCRIPTION:
This single-arm study aims to enroll 28 patients with unresectable malignant peritoneal mesothelioma. Enrolled patients will undergo treatment with sintilimab (200 mg), bevacizumab (7.5 mg/kg), pemetrexed (500 mg/m^2), and cisplatin (75 mg/m^2) administered every three weeks. Tumor assessments will be performed every two cycles according to RECIST 1.1 criteria, and after six cycles, maintenance therapy with sintilimab, bevacizumab, and pemetrexed will continue until disease progression or unacceptable toxicity occurs. The primary outcome measure of the study is Progression-Free Survival (PFS), while secondary outcomes include Overall Survival (OS), Objective Response Rate (ORR), and Disease Control Rate (DCR).

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and voluntarily sign the informed consent form;
2. Age ≥18 years old;
3. Pathologically (including histologically or cytologically) confirmed as peritoneal mesothelioma;
4. ECOG performance status of 0-1;
5. Expected survival of ≥3 months;
6. Function of vital organs must meet the following criteria (use of any blood products and cell growth factors is not allowed within 14 days prior to enrollment): Absolute neutrophil count ≥1.5×10^9/L; Platelets ≥100×10^9/L; Hemoglobin ≥90g/L; Total bilirubin <1.5 times the upper limit of normal (ULN); ALT and AST <2.5×ULN, GPT ≤1.5×ULN; Serum creatinine ≤1×ULN; Creatinine clearance rate >60 ml/min (Cockcroft-Gault formula);
7. Women of childbearing potential must have a negative serum pregnancy test within 7 days before enrollment and agree to use appropriate contraception during the trial and for 8 weeks after the last dose of trial medication; for men, must be surgically sterilized or agree to use appropriate contraception during the trial and for 8 weeks after the last dose of trial medication;
8. Have not participated in other clinical studies within 4 weeks before enrollment and during treatment. -

Exclusion Criteria:

1. Unable to adhere to the study protocol or procedures;
2. Vaccination with live vaccines within 4 weeks before enrollment or expected during the study period;
3. Other malignancies within the past 5 years, except for cured basal or squamous cell skin cancer, thyroid papillary carcinoma, or in situ cervical cancer;
4. Active autoimmune diseases or a history of autoimmune diseases within 4 weeks prior to enrollment;
5. Previous allogeneic bone marrow or organ transplantation;
6. Serious cardiovascular diseases within 6 months prior to enrollment, including unstable angina or myocardial infarction;
7. Allergy to study drugs or any of their excipients;
8. International Normalized Ratio (INR) >1.5 or Partial Thromboplastin Time (APTT) >1.5×ULN;
9. Electrolyte abnormalities of clinical significance as judged by the investigator;
10. Uncontrolled hypertension before enrollment, defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
11. Evidence or history of significant bleeding tendency within 3 months before enrollment (bleeding >30 mL, including hematemesis, melena, hematochezia), hemoptysis (more than 5 mL of fresh blood within 4 weeks) or a thromboembolic event (including stroke and/or transient ischemic attack) within the past 12 months;
12. Significant cardiovascular diseases of clinical importance, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within the past 6 months; congestive heart failure New York Heart Association (NYHA) class >2; ventricular arrhythmias requiring medication; Left Ventricular Ejection Fraction (LVEF) <50%;
13. Active or uncontrolled severe infections (≥CTCAE v5.0 Grade 2);
14. Known Human Immunodeficiency Virus (HIV) infection. Clinically significant liver disease history, including viral hepatitis [active Hepatitis B Virus (HBV) infection must be excluded, i.e., HBV DNA positive (>1×10^4 copies/mL or >2000 IU/mL); known Hepatitis C Virus (HCV) infection and HCV RNA positive (>1×10^3 copies/mL)];
15. Any other diseases, clinically significant metabolic dysfunctions, physical examination findings, or laboratory findings that, in the judgment of the investigator, make the patient unsuitable for the study drug (e.g., requiring treatment for epilepsy), could interfere with the interpretation of study results, or place the patient at high risk;
16. Urinalysis indicating urine protein ≥2+ and 24-hour urine protein >1.0g;
17. Complications requiring long-term treatment with immunosuppressants or systemic or local use of immunosuppressive corticosteroids (more than 10mg/day of prednisone or equivalent therapeutic hormones);
18. Patients deemed unsuitable for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 36 months
  The time from the date of first administration of this regimen to the date of first documented disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 36 months
  The time from the initiation of the first dose of medication in a patient to death from any cause.
Objective Response Rate (ORR) | 36 months
  The proportion of patients with a comfirmed complete response or patial response using RECIST1.1.
Disease Control Rate (DCR) | 36 months
  The percentage of patients who have achieved complete response, partial response, and stable disease to the treatment, as defined by RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Yongkun Sun, Doctor, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical SciencesCancer
Locations (1):
- Cancer Institute and Hospital,Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No